CLINICAL TRIAL: NCT07365826
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Clinical Study to Evaluate the Safety, Tolerability, and Immunogenicity of VAX-31 Concomitantly Administered With Seasonal Influenza Vaccine in Healthy Subjects 50 Years of Age and Older
Brief Title: A Clinical Study to Evaluate the Safety, Tolerability, and Immunogenicity of VAX-31 With Influenza Vaccine in Adults ≥ 50 Years of Age
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vaxcyte, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VAX31-106
Record Dates: First submitted 2026-01-22; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Pneumococcal Vaccines
Keywords: 31-Valent PCV; Pneumonia; Pneumococcal Infection
MeSH Terms: conditions — Pneumonia; Pneumococcal Infections | interventions — FluBlok

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VAX-31 + SIV (Experimental): Participants will receive a single dose of VAX-31 administered as an intramuscular injection at Day 1, concomitantly administered with SIV, followed by placebo at Month 1.
  Interventions: Biological: 31-valent pneumococcal conjugate vaccine; Biological: Seasonal Influenza Vaccine (SIV) (Flublok); Biological: Placebo
- Placebo + SIV (Experimental): Participants will receive placebo administered via intramuscular injection at Day 1, concomitantly administered with SIV, followed by VAX-31 at Month 1.
  Interventions: Biological: 31-valent pneumococcal conjugate vaccine; Biological: Seasonal Influenza Vaccine (SIV) (Flublok); Biological: Placebo

INTERVENTIONS:
Biological: 31-valent pneumococcal conjugate vaccine — 0.5 mL of VAX-31 will be administered into the deltoid muscle
Biological: Seasonal Influenza Vaccine (SIV) (Flublok) — 0.5 mL of SIV into the deltoid muscle
Biological: Placebo — 0.5mL of placebo (normal saline) into the deltoid muscle

SUMMARY:
This is a Phase 3, randomized, double-blind study to evaluate the safety and immunogenicity of VAX-31 and seasonal influenza vaccine in pneumococcal-naïve adults ≥ 50 years when the two vaccines are administered at the same visit or separately.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥50 years of age (inclusive) at the time of randomization into the study.
2. Able and willing to complete the informed consent process.
3. Available for clinical follow-up through the last study visit at 7 months after the first study vaccination.
4. In good general health or with stable underlying chronic condition(s), as determined by medical history, oral temperature, physical examination, and clinical judgment of the Investigator.
5. Willing to have blood samples collected and used for research purposes.
6. Able to provide proof of identity to the satisfaction of the study site personnel completing the enrollment process.
7. Female subjects of childbearing potential, defined as premenopausal females capable of becoming pregnant, must have a negative urine pregnancy test at Screening and immediately prior to each vaccination and agree to use acceptable contraception, if heterosexually active. Female subjects who are not abstinent from heterosexual intercourse must agree to consistently practice contraception at least 7 days prior to vaccination and through their last study visit. Male subjects with partners of childbearing potential must agree to practice an acceptable contraception method ([use condoms with or without spermicide] or have undergone a vasectomy) from Day 1 through their last study visit. Note: A history of amenorrhea for at least 12 months without an alternative medical cause is required for a female to be considered postmenopausal in the study.
8. Able to access and use a device connected to Wi-Fi or cellular network for completion of an electronic diary (eDiary).

Exclusion Criteria:

1. History of IPD or pneumococcal pneumonia (either confirmed or self-reported) at any age.
2. Previous receipt of a licensed or investigational pneumococcal vaccine at any age.
3. Previous receipt of an influenza vaccine from the current season; receipt of any influenza vaccine (licensed or investigational) within 6 months prior to Day 1; or receipt/planned receipt of any licensed or investigational non-study influenza vaccine during study participation.
4. Receipt of any investigational product within 30 days prior to Day 1, currently participating in another interventional investigational study, or having plans to receive another investigational product(s) while on study.
5. Planned or actual administration of any licensed vaccine within 30 days prior to Day 1.
6. Body temperature >38.0°C (>100.4°F) or acute illness within 3 days prior to study vaccination (participant may be rescreened).
7. Current diagnosis of human immunodeficiency virus (HIV), Hepatitis B, or Hepatitis C.
8. History of severe allergic reaction with generalized urticaria, angioedema, or anaphylaxis to any previous vaccination.
9. History of Guillain-Barré syndrome.
10. Individual who is pregnant, breastfeeding, or planning to become pregnant during study participation.
11. Has a known or suspected immunocompromising condition, including, but not limited to, leukemia, lymphoma, chronic renal failure, or congenital or acquired immunodeficiency.
12. Bleeding disorder diagnosed by a doctor (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions) resulting in clinically significant bruising or bleeding difficulties with IM injections or blood draws.
13. Receipt of blood or blood product (including polyclonal intravenous immunoglobulin) within 60 days prior to Day 1.
14. Receiving immunosuppressive therapy.
15. Received any part of a ≥14-day course of systemic corticosteroids (prednisone equivalent >10 mg/day) within 14 days of study vaccinations. Note: Receipt of a ≥14-day course of systemic corticosteroids equivalent to ≤10 mg/day is permitted, as are inhaled, nebulized, topical, intra-articular, and intrabursal corticosteroids.
16. History of malignancy ≤5 years before to Day 1, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer.
17. Any medical, psychiatric, or social condition that in the judgment of the Investigator is a contraindication to protocol participation or impairs a participant's ability to give informed consent.
18. Employee of, or first-degree relative of any person employed by the Sponsor, the contract research organization (CRO), the Investigator, study site personnel, or site.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
For each of the 32 serotypes (the 31 serotypes included in VAX-31, and serotype 20B), the ratio (co-administration group to sequential administration group) of opsonophagocytic activity (OPA) geometric mean titers (GMT) in evaluable participants | 1 Month after VAX-31 vaccination
For each of the strains in SIV, the ratio (co-administration group to sequential administration group) of hemagglutination inhibition (HAI) GMT in evaluable participants | 1 Month after SIV administration
Percentage of participants reporting solicited local adverse events (AE) within 7 days after Day 1 and Month 1 vaccination (redness, swelling, and pain at injection site) in each group | 7 days after each vaccination
Percentage of participants reporting solicited systemic AE within 7 days after Day 1 and Month 1 vaccination (fever, headache, fatigue, muscle pain, and joint pain) in each group | 7 days after each vaccination
Percentage of participants reporting unsolicited AE within 1 month after Day 1 and Month 1 vaccination in each group | 7 days after each vaccination
Percentage of participants reporting NOCI, MAAE, and SAE within 6 months after last vaccination in each group | 6 Months after last vaccination

SECONDARY OUTCOMES:
For each of the 32 serotypes (the 31 serotypes included in VAX-31, and serotype 20B), the ratio (co-administration group to sequential administration group) of IgG geometric mean concentrations (GMC) in evaluable participants | 1 month after VAX-31 administration

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - Hope Research Institute, Phoenix, Arizona
  - Tekton Research at Fort Collins, Fort Collins, Colorado
  - University Clinical Research - Deland, DeLand, Florida
  - CenExel Research Centers of America, Hollywood, Florida
  - Health Awareness, Jupiter, Florida
  - Accel Research Sites - Lakeland, Lakeland, Florida
  - Accel Research Sites - Largo, Largo, Florida
  - Precision Clinical Research, Sunrise, Florida
  - Velocity Valparaiso, Valparaiso, Indiana
  - Johnson County ClinTrials, Lenexa, Kansas
  - AMR Lexington, Lexington, Kentucky
  - DM Clinical Research - Detroit, Detroit, Michigan
  - Velocity Omaha, Omaha, Nebraska
  - Rochester Clinical Research, Rochester, New York
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - DelRicht Research - Hendersonville, Hendersonville, Tennessee
  - AMR Knxoville, Knoxville, Tennessee
  - Tekton Research at Austin, Austin, Texas
  - REX Clinical Trials, Beaumont, Texas
  - Epic Medical Research, DeSoto, Texas
  - CenExel JBR Clinical Research, Salt Lake City, Utah
  - Charlottesville Medical Research Center, Charlottesville, Virginia
  - Health Research of Hampton Roads, Inc., Newport News, Virginia
  - Clinical Research Partners, LLC., Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Vaxcyte is committed to providing access to anonymized data from the company's clinical trials for the purpose of legitimate scientific research. Requests for data may be addressed to datasharing@vaxcyte.com. Requests must be accompanied by a detailed analysis plan and will be reviewed for scientific validity. Data will be made available after initial product approval. Sharing of data may require execution of a data-sharing agreement.
Supporting Information: Study Protocol
Time Frame: Individual participant data will be shared after deidentification and made available starting 6 months after initial product approval.
Access Criteria: Criteria will depend on the specific proposal received and may include qualification of the scientific researchers, potential contribution to the research field, scientific rigor of statistical and analytical methods, and other criteria appropriate for the proposal.